CLINICAL TRIAL: NCT03369665
Title: A 2-Year Prospective Study to Assess Health-related Quality of Life In Subjects With Highly-Active Relapsing Multiple Sclerosis Treated With Mavenclad® (CLARIFY MS)
Brief Title: Evaluation of Quality of Life (QoL) in Subjects With Highly Active Relapsing Multiple Sclerosis (MS) (CLARIFY MS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS700568_0021; 2017-002632-17 (EudraCT Number)
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Mavenclad®; Cladribine; Health-related Quality of Life
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mavenclad® (Experimental)
  Interventions: Drug: Mavenclad®

INTERVENTIONS:
Drug: Mavenclad® — Participants with Relapsing Multiple Sclerosis (RMS) received Mavenclad® 3.5 milligram per kilogram (mg/kg) of body weight over 2 years, administered as 1 treatment course of 1.75 mg/kg per year. Each treatment course consisted of 2 treatment weeks, one at the beginning of the first month and one at the beginning of the second month of the respective year.
  Other Names: Cladribine

SUMMARY:
The main purpose of the study was to assess the health-related quality of life (HRQoL) through the Multiple Sclerosis Quality of Life-54 Questionnaire (MSQoL-54) scale in highly-active relapsing multiple sclerosis (RMS) particpants treated with Mavenclad® for 2 years (24 months).

ELIGIBILITY:
Inclusion Criteria:

* Highly active RMS as defined by:
* One relapse in the previous year and at least 1 T1 Gadolinium (Gd)+ lesion or 9 or more T2 lesions, while on therapy with other disease modifying drugs (DMDs).
* Two or more relapses in the previous year, whether on DMD treatment or not.
* Expanded Disability Status Scale (EDSS) score less than equals to (<=) 5.0.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Positive hepatitis C or hepatitis B surface antigen test and/or core antibody test for immunoglobulin G (IgG) and/or immunoglobulin M (IgM).
* Current or previous history of immune deficiency disorders including a positive human immunodeficiency virus (HIV) result.
* Currently receiving immunosuppressive or myelosuppressive therapy with, for example, monoclonal antibodies, methotrexate, cyclophosphamide, cyclosporine or azathioprine, or chronic use of corticosteroids.
* History of tuberculosis, presence of active tuberculosis, or latent tuberculosis
* Presence of Progressive Multifocal Leukoencephalopathy (PML) in Magnetic Resonance Imaging (MRI).
* Active malignancy.
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (90):
- Austria (3):
  - Kepler Universitätsklinikum, Linz
  - Paracelsus Medical University Salzburg, Salzburg
  - Eva Maida, Vienna
- Belgium (3):
  - Cliniques Univ. St.-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Clinique Saint Pierre, Ottignies
- Czechia (8):
  - FN u sv. Anny Brno, Brno
  - FN Hradec Kralove, Choceň
  - Nemocnice Jihlava, p.o., Jihlava
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava (11573), Ostrava
  - Faculty Hospital Kralovske Vinohrad, Prague
  - Vseobecna fakultni nemocnice v Praze (11163), Prague
  - Nemocnice Teplice, Teplice
- Denmark (4):
  - Aalborg Hospital, Aalborg
  - Glostrup University Hospital, Glostrup Municipality
  - Odense Univeristy Hospital, Odense
  - Matthias Kant, Sønderborg
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Terveystalo Mikkeli, Mikkeli
  - Neo Research, Neuro NEO Oy, Turku
- France (13):
  - Centre hospitalier de la Côte Basque - Saint Léon, Bayonne
  - Hopital Pellegrin, Bordeaux
  - University Hospital of Caen, Caen
  - CHRU de Lille, Lille
  - Groupe Hospitalier de l'Institut Catholique de Lille - Centre Hospitalier Saint Philibert, Lomme
  - CHU de Nantes, Nantes
  - Centre Hospitalier de Gonesse, Paris
  - Hôpital de la Pitié-Salpétrière, Paris
  - CHU de Poissy, Poissy
  - CHU Hopital Gabriel Montpied, Puy-de-Dome
  - Centre Universitaire de Rouen, Rouen
  - Hopital Pierre-Paul Riquet - Neurologie, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
- Greece (3):
  - Hos. Errikos Dynan, Athens
  - 401 Army Hospital, Athens
  - Athens Medical Centre, Athens
- Hungary (6):
  - Semmelweis Egyetem AOK, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Jahn Ferenc Dél-Pesti Kórház és Rendelőintézet, Budapest
  - University of Debrecen, Debrecen
  - VALEOMED Kft, Esztergom
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór, Nyíregyháza
- Italy (13):
  - A.O.U. Ospedali Riuniti Umberto I, Ancona
  - Ospedale Binaghi, Università di Cagliari,ASL 8 - Centro Sclerosi Multipla, Cagliari
  - Policlinico di Catania, Catania
  - Ospedale San Raffaele Giglio, Cefalù
  - Ospedale San Raffaele, IRCCS, Milan
  - Instituto Nazionale Neurologico "Carlo Besta", Milan
  - A.O. Universitaria Federico II, Napoli
  - Seconda Univesità degli Studi di Napoli, AOU, Napoli
  - Villa Sofia Hospital, Palermo
  - Azienda Ospedaliera S. Camillo Forlanini (8025), Roma
  - Azienda Ospedaliera Sant'Andrea Università La Sapienza, Roma
  - Neurological Center Of Latium, Roma
  - Policlinico Tor Vergata, Roma
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Klaipedos Ligonine, Kaunas
  - Vilnius University Hospital Santariskiu Clinics, Vilnius
- Zuyderland, Sittard-Geleen, Netherlands
- Drammen Hospital, Drammen, Norway
- Poland (7):
  - COPERNICUS Podmiot Leczn. Sp z o.o., Gdansk
  - M.A. - LEK A.M.Maciejowscy SC., Katowice
  - Centrum Neurologii K. Selmaj, Lodz
  - Uniwersytecki Szpital Kliniczny nr 1 i.m. Norberta Barlickie, Lodz
  - Centrum Medyczne Medyk, Lublin
  - Indywidualna Praktyka Lekarska Prof. Konrad Rejdak, Lublin
  - Instytut Psychiatrii i Neurologii, Warsaw
- Portugal (2):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Porto E.P.E. Hospital de Santo António, Porto
- Slovakia (4):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica Nitra, Nitra
  - Fakultna nemocnica Trnava, Trnava
- Spain (10):
  - C.A.U. de León - H. de León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón (5030), Madrid
  - H. U. Quirónsalud Madrid, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí
  - Hospital Universitario Nuestra Senora de la Candelaria (4776), Santa Cruz de Tenerfie
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio - Servicio de Oncologia, Seville
- Sweden (2):
  - Karlstad Hospital (8232), Karlstad
  - Motala Hospital (11119), Motala
- United Kingdom (4):
  - Institute of Neurological Sciences, Glasgow
  - GM LCRN - Great Manchester Local Clinical Research Network, Manchester
  - The Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Morriston Hospital (4232), Swansea West Glamorgan

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] Brochet B, Solari A, Lechner-Scott J, Piehl F, Langdon D, Hupperts R, Selmaj K, Patti F, Brieva L, Maida EM, Alexandri N, Smyk A, Nolting A, Keller B, Montalban X, Kubala Havrdova E. Improvements in quality of life over 2 years with cladribine tablets in people with relapsing multiple sclerosis: The CLARIFY-MS study. Mult Scler. 2023 Dec;29(14):1808-1818. doi: 10.1177/13524585231205962. Epub 2023 Nov 18. PMID 37978852
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0021
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 485 participants were enrolled in the study from different trial sites across Poland, Czechia, Slovakia, Hungary, Lithuania, Austria, Denmark, Finland, Sweden, Norway, Italy, Spain, Portugal, Greece, France, Netherlands, United Kingdom of Great Britain and Northern Ireland, and Belgium. Out of 485 participants, three participants were enrolled, but did not receive study medication.
Period: Overall Study
Arm/Group | Mavenclad®
Started | 482
Full Analysis Set (FAS) (Full Analysis Set (FAS) consisted of all participants from the Intent-to-treat (ITT [ITT population included all participants classified as eligible]) set treated with at least one dose of study medication.) | 482
Safety Analysis Set (SAS) (SAF consisted of all participants treated with at least one dose of study medication.) | 482
Completed | 452
Not Completed | 30
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 15
Not completed — Progression Disease | 2
Not completed — Not classified | 3

BASELINE CHARACTERISTICS:
Population: FAS consisted of all participants from the ITT set treated with at least one dose of study medication.
Arm/Group | Mavenclad®
Number analyzed (Participants) | 482
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.4 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 338
  Male | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 379
  Unknown or Not Reported | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 360
  Race: Asian | 2
  Race: Not collected at this site | 120

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Multiple Sclerosis Quality of Life-54 Questionnaire (MSQoL-54) Physical Health Composite Summary and Mental Health Composite Summary Scores at Month 24
Description: The MSQOL-54 was a multidimensional health-related QOL measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 sub-scales along with two summary scores, and two additional single-item measures. Sub-scales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The two summary scores physical health and mental health are derived from a weighted combination of scale scores. Each composite summary score has a range from 0-100 where higher scores indicate better QOL. A positive change from baseline indicates improvement.
Time Frame: Baseline, Month 24
Population: FAS consisted of all participants from the ITT set treated with at least one dose of study medication. Here, "overall number of participants analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Mavenclad®
Number analyzed (Participants) | 433
Score on a Scale
  Physical health composite summary | 4.86 (0.769)
  Mental health composite summary | 4.80 (0.845)

2. Secondary Outcome: Treatment Global Satisfaction Determined by Treatment Satisfaction Questionnaire Medication Version 1.4 (TSQM v1.4) Scale at Month 6
Description: TSQM version 1.4 was a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. It comprises of 14 items assessing the following 4 domains: effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions:12-14). Global Satisfaction- Question 12 scored as 1 (not at all confident) to 5 (extremely confident); question 13 scored as 1 (not at all certain) to 5 (extremely certain); and question 14 scored as 1 (extremely dissatisfied) to 7 (extremely satisfied). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction.
Time Frame: At Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Mavenclad®
Number analyzed (Participants) | 477
Score on a Scale | 72.02 (1.528)

ADVERSE EVENTS:
Time Frame: From Baseline up to Month 24
Description: Safety Analysis Set (SAF) consisted of all participants treated with at least one dose of study medication.
Arm/Group | Mavenclad®
All-Cause Mortality (participants affected / at risk) | 0/482
Serious Adverse Events (participants affected / at risk) | 26/482
Other Adverse Events (participants affected / at risk) | 375/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavenclad® (N=482)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 1
Lyme disease (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Medication error (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Ovulation pain (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavenclad® (N=482)
Lymphopenia (Blood and lymphatic system disorders) | 73
Nausea (Gastrointestinal disorders) | 25
Fatigue (General disorders) | 30
Influenza (Infections and infestations) | 29
Nasopharyngitis (Infections and infestations) | 65
Oral herpes (Infections and infestations) | 25
Upper respiratory tract infection (Infections and infestations) | 47
Urinary tract infection (Infections and infestations) | 39
Back pain (Musculoskeletal and connective tissue disorders) | 38
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26
Headache (Nervous system disorders) | 105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03369665/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03369665/SAP_001.pdf